CLINICAL TRIAL: NCT06261190
Title: Study Protocol of Extended Multicenter Prospective Cohort Study of Active Surveillance on Papillary Thyroid Carcinoma (MAeSTro-EXP)
Brief Title: Active Surveillance for Low-risk Papillary Thyroid Carcinoma
Acronym: MAeSTro-EXP
Status: Enrolling by invitation | Type: Observational
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other); Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-2308-182-1463
Record Dates: First submitted 2024-01-25; First posted 2024-02-15 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Thyroid Cancer; Papillary Thyroid Carcinoma
Keywords: Active Surveillance; Immediate surgery
MeSH Terms: conditions — Thyroid Neoplasms; Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Active surveillance: Group with active surveillance of their Papillary Thyroid Cancer
- Immediate surgery: Group who underwent surgery after diagnosis Papillary Thyroid Cancer

SUMMARY:
This is a multi-center, non-randomized, prospective observational cohort study aimed at establishing a cohort of low-risk papillary thyroid cancer patients with a maximum tumor diameter of 1.5 cm or less, consisting of an active surveillance group and an immediate surgery group.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the natural course of low-risk papillary thyroid cancer, specifically the progression rates of tumor size increase and the occurrence of local or distant metastasis. Ultimately, it is expected that establishing new criteria for active surveillance of low-risk papillary thyroid cancer in Korean patients will lead to a reduction in unnecessary surgical treatments, improving quality of life and decreasing national healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* subjects over 18 years old with a thyroid nodule of ≤ 1.5 cm in maximum diameter and a Bethesda category V or VI diagnosis on cytopathology
* subjects without high-risk features, including lymph node (LN) metastasis, distant metastasis, signs or symptoms of invasion to the recurrent laryngeal nerve or trachea, Poorly differentiated cancer or variant with a poor prognosis, such as the tall cell, diffuse sclerosing, columnar cell, or solid variants.

Exclusion Criteria:

* subjects who are unable or unwilling to attend regular follow-ups..
* subjects with a diagnosis of benign, atypia of undetermined significance, suspicious for follicular neoplasm, or follicular neoplasm (Bethesda category II, III, or IV) based on Fine needle aspiration or, or benign, indeterminate by core needle biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects aged older than 18 years with the tumor size of ≤ 1.5 cm papillary thyroid carcinoma, who meet the inclusion criteria from Seoul National University Hospital, National Cancer Center, Seoul National University Bundang Hospital, and SMG-SNU Boramae Medical Center.
Sampling Method: Probability Sample
Enrollment: 499 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of disease progression between the active surveillance group and the immediate surgery group | At 5years, 10years after enrollment
  Disease progression in the following criteria: (1) a size increase of ≥3 mm in maximum diameter or size increase of ≥2 mm in two diameters; (2) a cytopathological diagnosis of a new thyroid cancer lesion; (3) a cytopathological diagnosis of a cervical lymph node metastasis; or (4) clinical or radiological suspicion of a distant metastasis.

SECONDARY OUTCOMES:
Risk factors for disease progression in the active surveillance group | At 5years, 10years after enrollment
  To evaluate the risk factors for progression to thyroid cancer based on demographic factors, serial ultrasound findings, blood markers, and molecular pathological characteristics at each follow-up visit.
Rate of conversion to surgery without disease progression in the active surveillance group | At 5years, 10years after enrollment
  To estimate the proportion of patients in the active surveillance group who undergo surgery without clinical evidence of progression to thyroid cancer, evaluated at each follow-up visit.
Rate of Disease Progression Between the Immediate Surgery Group and the Surgery-After-Progression Group | At 5years, 10years after enrollment
  The outcome will be measured as the proportion (%) of patients in each group who experience disease progression at each follow-up visit.
  Disease progression is defined as meeting any of the following criteria:
  1. an increase in tumor size of ≥3 mm in maximum diameter, or ≥2 mm in two perpendicular diameters;
  2. a cytopathological diagnosis of a new thyroid cancer lesion;
  3. a cytopathological diagnosis of cervical lymph node metastasis;
  4. clinical or radiological suspicion of distant metastasis.
Factors influencing treatment decision-making | At 5years, 10years after enrollment
  To evaluate the factors influencing the decision to pursue active surveillance, undergo surgery, or modify the treatment.
Decision Conflict Scale Score | For the first 2 years, every 6 months, then every 6-12 months depending on the condition.
  The level of confidence in decision-making will be assessed at each follow-up visit using the Decision Conflict Scale. This questionnaire evaluates the level of agreement with statements related to treatment plan decisions on a scale from 0 (strongly disagree) to 5 (strongly agree), in 1-point increments. Higher scores indicate greater confidence and certainty in the decision-making process.
Shared Decision-Making Satisfaction Score | For the first 2 years, every 6 months, then every 6-12 months depending on the condition.
  To assess patient satisfaction with the shared decision-making process with healthcare providers. Satisfaction is measured using a questionnaire rated on a scale from 0 (very dissatisfied) to 10 (very satisfied), with 1-point increments. Higher scores indicate greater satisfaction with the collaborative decision-making process.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - SMC-SNU Boramae Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: Undecided